CLINICAL TRIAL: NCT01578850
Title: A Randomized, Double-blind Placebo-controlled Study Of The Maintenance Of Efficacy Of Etanercept Plus Dmard(s) Compared With Dmard(s) Alone In Subjects With Rheumatoid Arthritis After Achieving An Adequate Response With Etanercept Plus Dmard(s)
Brief Title: Study Conducted in Subjects With Rheumatoid Arthritis Who Have Moderate to Severe Disease Activity Despite Methotrexate Therapy With or Without Other Non Biologic Disease Modifying Antirheumatic Drugs (DMARDs)for at Least 12 Weeks Prior to Screening
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1801315; 2011-005448-87 (EudraCT Number); B1801315 (Other: Alias Study Number)
Record Dates: First submitted 2012-04-12; First posted 2012-04-17 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-05

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; etanercept; methotrexate; DMARDs
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: Etanercept
- Group B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Etanercept — etanercept 50mg once weekly + methotrexate with or without other DMARDs
  Arms: Group A
Drug: placebo — etanercept placebo once weekly + methotrexate with or without other DMARDs
  Arms: Group B

SUMMARY:
To compare the maintenance of efficacy of the combination of etanercept 50 mg once weekly plus methotrexate with or without other disease modifying antirheumatic drugs therapy with that of methotrexate with or without other disease modifying antirheumatic drugs therapy at Week 52 in subjects with moderately to severely active rheumatoid arthritis who have achieved low disease activity after 24 weeks of therapy with open label etanercept 50 mg once weekly plus MTX with or without other disease modifying antirheumatic drugs therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has a minimum 1 year history/diagnosis of rheumatoid arthritis based on the 1987 American College of Rheumatology (ACR) Revised criteria for RA.
2. Subject must have active rheumatoid arthritis despite methotrexate (MTX) therapy of ≥10 mg/wk for at least 12 weeks. The MTX dose must be stable for at least 4 weeks immediately prior to screening.

Exclusion Criteria:

1. Subjects who used any of the following systemic treatments during the washout periods given below:

   1. Oral corticosteroid dose of prednisone >7.5 mg/day (or equivalent) or a change in dose within 28 days of baseline.
   2. Treatment with more than 1 NSAID within 14 days at baseline.
   3. Methotrexate dose greater than 25 mg/week, or change in the dose of methotrexate within 28 days of baseline.
   4. Subjects will be allowed to continue the following non biologic DMARDs: sulfasalazine, hydroxychloroquine, and leflumomide. All other non-biologic DMARDs (including but not limited to gold, penicillamine, azathioprine, cyclophospamide), and biologic DMARDs must have been discontinued at least 2 months prior to Week 1.
   5. Any biologic B cell depleting agent (eg, rituximab) within 2 years of Week 1.
2. Receipt of any live (attenuated) vaccine within 4 weeks prior to baseline.
3. Receipt of any live (attenuated) vaccine within 4 weeks prior to baseline.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (62):
- Brazil (4):
  - Hospital Santa Izabel - Santa Casa de Misericórdia da Bahia, Salvador, Estado de Bahia
  - CIP (Centro Internacional de Pesquisa), Goiânia, Goiás
  - CEPIC - Centro Paulista de Investigacao Clinica e Servicos Medicos LTDA, São Paulo, São Paulo
  - Research Center, Juiz de Fora
- China (4):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Chinese Academy of Medical Sciences - Peking Union Medical C, Beijing
  - Shanghai Changning District Guanghua Hospital of Traditional Chinese and Western Medicine, Shanghai
  - Shanghai Changhai Hospital[Rheumatology &Immunology], Shanghai
- Colombia (3):
  - Hospital Pablo Tobon Uribe (HPTU), Santa Fe de Antioquia, Antioquia
  - Centro Integral de reumatolo[Gerencia / Representante Legal], Barranquilla, Atlántico
  - Fundacion Instituto de Reumatologia Fernando Chalem, Bogota DC, Cundinamarca
- Czechia (4):
  - Revmatologicka poradna III. Interni nefrologicka, revmatologicka a endokrinologicka klinika, Olomouc, Czech Republic
  - Revmatologicky ustav, Prague, Czech Republic
  - Revmatologicka ambulance, Prague, Czech Republic
  - PV-Medical s.r.o., Zlín, Czech Republic
- Egypt (3):
  - New University Hospital, Alexandria Clinical Research Center, Alexandria, Alexandria Governorate
  - Al Azhar University Hospital [Rheumatology], Cairo, Cairo Governorate
  - Ain Shams University/Al Demerdash Hospital/Diabetology Unit, Cairo
- Hungary (2):
  - Budai Irgalmasrendi Korhaz, Budapest
  - Magyar Honvédség Egészségügyi Központ, Budapest
- Pharmaceutical Research Center- PRC. Jordan University of Science and Technology, Irbid, Jordan
- American University of Beirut Medical Center, Beirut, Lebanon, Lebanon
- Malaysia (3):
  - Hopsital Putrajaya [Medicine], Putrajaya, Putrajaya
  - Queen Elizabeth Hospital, Kota Kinabalu, Sabah
  - University Malaysia Medical Centre, Kuala Lumpur
- Mexico (4):
  - Centro de Investigación y Atención Integral de Durango, SC, Durango, Durango / Mexico
  - Centro de Alta Especialidad en Reumatología e Investigación, San Luis de Potosi, San Luis Potosí / Mexico
  - Centro Medico Las Americas, Mérida, Yucatán
  - Hospital Central, San Luis Potosí City
- Philippines (5):
  - De La Salle University Health Sciences Campus- Clinical Epidemiology Unit, Dasmariñas, Cavite
  - St. Luke's Mecical Center, Quezon, Manila
  - Angeles University Foundation Medical Center, Angeles City, Pampanga
  - Chong Hua Hospital, Medical Arts Center, Cebu City
  - UP-Philippine General Hospital, Medical Research Laboratory, Medicine Department,, Manila
- Hamad Medical Corporation, Doha, Qatar, Qatar
- Romania (4):
  - Spitalul Clinic Judetean de Urgenta Brasov, Brasov, Brașov County
  - Spitalul Clinic de Recuperare, Iași, Iaşi
  - Spitalul Judetean, Baia Mare, Maramure
  - Spitalul Clinic Judetean de Urgenta Targu Mures, Tg Mures
- Russia (6):
  - LLC Research Medical Complex Your Health based on City Clinical Hospital Number 7(Legal address), Kazan'
  - LLC Research Medical Complex Your Health based on City Clinical Hospital Number 7 (Actual address), Kazan'
  - Krasnoyarsk State Medical University named after Professor V.F. Voyno-Yasenetsky, Krasnoyarsk
  - Krasnoyarsk State Medical University named after Professor V.F. Voyno-Yasenetsky,, Krasnoyarsk
  - FSBSI "Scientific Research Institute of Rheumatology n. a. V.A. Nasonova", Moscow
  - LLC Institute of Medical Trials (Actual address), Saint Petersburg
- South Africa (3):
  - Universitas Hospital [Cardiololgy], Bloemfontein, Free State
  - Vincent Pallotti Hospital, Cape Town
  - Winelands Medical Research Centre, Stellenbosch
- Taiwan (4):
  - Cathay General Hospital, Dawan, Taoyuan
  - Buddhist Tzu Chi General Hospital - Dalin Branch, Chiayi City
  - China Medical University Hospital, Division of Rheumatology, Allergy and Immunology, Taichung
  - Taipei Medical University Hospital, Taipei
- Thailand (4):
  - Division of Rheumatology, Department of Internal Medicine, Faculty of Medicine,, Amphoe Mueang, Chiang Mai
  - Siriraj Hospital [Rheumatology], Bangkok
  - Khon Kaen University (KKU) - Faculty of Medicine, Khon Kaen
  - Songklanagarind Hospital, Songkhla
- Ukraine (5):
  - Republican Clinical Hospital, Department of Internal Medicine #2 of Crimean State Medical University, Simferopol, Autonomous Republic of Crimea
  - Komunalnyi zaklad Kyivskoi oblasnoi rady "Kyivska oblasna klinichna likarnia", Kyiv
  - Odessa Regional Clinical Hospital, Outpatient Department, Odesa
  - Municipal Institution of Ternopil Regional Council Ternopil University Hospital, Ternopil
  - Vinnitsa Regional Clinical Hospital n.a. Pirogov, Department of Faculty Therapy of Vinnitsa NMU, Vinnitsa
- Al Baraha Hospital, Dubai, United Arab Emirates

REFERENCES:
- [Derived] Tanaka Y, Smolen JS, Jones H, Szumski A, Marshall L, Emery P. The effect of deep or sustained remission on maintenance of remission after dose reduction or withdrawal of etanercept in patients with rheumatoid arthritis. Arthritis Res Ther. 2019 Jul 5;21(1):164. doi: 10.1186/s13075-019-1937-4. PMID 31277720
- [Derived] Zerbini CAF, Abud-Mendoza C, Mendez-Patarroyo P, De Angelo Andrade M, Pedersen R, Vlahos B, Borlenghi CE. Maintenance of low disease activity and remission with etanercept-disease-modifying antirheumatic drug (DMARD) combination therapy compared with treatment with DMARDs alone in Latin American patients with active rheumatoid arthritis: Subset analysis of a randomized trial. Medicine (Baltimore). 2018 Sep;97(36):e11989. doi: 10.1097/MD.0000000000011989. PMID 30200078
- [Derived] Pavelka K, Akkoc N, Al-Maini M, Zerbini CAF, Karateev DE, Nasonov EL, Rahman MU, Pedersen R, Dinh A, Shen Q, Vasilescu R, Kotak S, Mahgoub E, Vlahos B. Maintenance of remission with combination etanercept-DMARD therapy versus DMARDs alone in active rheumatoid arthritis: results of an international treat-to-target study conducted in regions with limited biologic access. Rheumatol Int. 2017 Sep;37(9):1469-1479. doi: 10.1007/s00296-017-3749-7. Epub 2017 Jun 9. PMID 28597306
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1801315&StudyName=Study%20conducted%20in%20subjects%20with%20rheumatoid%20arthritis%20who%20have%20moderate%20to%20severe%20disease%20activity%20despite%20methotrexate%20therapy%20with%20or%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study consisted of Period 1 (an open-label, 24-week treat-to-target period), and Period 2 (a double-blind, randomized, 28-week period for participants who qualified for randomization).
Pre-assignment Details: The study was conducted in participants with rheumatoid arthritis (RA) who had moderate to severe disease activity despite methotrexate (MTX) therapy (≥10 mg/week) with or without other non-biologic disease modifying anti-rheumatic drugs (DMARDs) for at least 12 weeks prior to screening.
Groups:
- Open-Label Treatment: Participants in open-label treatment received Etanercept (ETN) 50 milligram (mg) once a week (QW) with MTX (with or without other DMARDs).
- Etanercept: Participants were randomized to receive ETN 50 mg QW with MTX (with or without other DMARDs).
- Placebo: Participants were randomized to receive PBO 50 mg QW + MTX (with or without DMARDs).
Period: Period 1
Arm/Group | Open-Label Treatment | Etanercept | Placebo
Started | 489 (491 participants were enrolled in open-label treatment but 2 did not receive study medication.) | 0 | 0
Completed | 452 | 0 | 0
Not Completed | 37 | 0 | 0
Not completed — Insufficient Clinical Response | 1 | 0 | 0
Not completed — Adverse Event | 11 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Does Not Meet Entrance Criteria | 12 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0
Not completed — Study Terminated by Sponsor | 3 | 0 | 0
Period: Period 2
Arm/Group | Open-Label Treatment | Etanercept | Placebo
Started | 0 | 167 (Two participants in ETN did not receive treatment.) | 176 (One participants in PBO did not receive treatment.)
Completed | 0 | 154 | 162
Not Completed | 0 | 13 | 14
Not completed — Insufficient Clinical Response | 0 | 1 | 0
Not completed — Adverse Event | 0 | 3 | 6
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 2
Not completed — Study Terminated by Sponsor | 0 | 5 | 4
Not completed — Unspecified Reasons | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set for Period 2 (Double Blind FAS) included all randomized participants who met the period 2 DAS28-ESR inclusion criteria, had at least one dose of study drug during Period 2 (ie, ETN, MTX or placebo) and have at least one valid efficacy (DAS28-ESR) evaluation after randomization.
Groups:
- Placebo: Participants were randomized to receive PBO 50 mg QW with MTX (with or without other DMARDs).
- Total: Total of all reporting groups
Arm/Group | Etanercept | Placebo | Total
Number analyzed (Participants) | 167 | 176 | 343
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.2 (12.88) | 47.0 (12.02) | 46.6 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 150 | 290
  Male | 27 | 26 | 53

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Remained in Low Disease Activity (LDA) (Disease Activity Score in 28 Joints-erythrocyte Sedimentation Rate [DAS28-ESR] <3.2) at Week 52.
Description: Proportion of participants who remained in LDA DAS28-ESR <3.2 at Week 52 is presented below.
Time Frame: Baseline and Week 52
Population: The FAS included all randomized participants who met the period 2 DAS28-ESR inclusion criteria, had at least one dose of study drug during Period 2 (ie, ETN, MTX or PBO) and had at least one valid efficacy (DAS28-ESR) evaluation after randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
percentage of participants | 43.6 | 17.3
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Stratified by geographic region and disease status at randomization (Stratum 1=Remission: DAS28-ESR<2.6 or Stratum 2=LDA: 2.6<=DAS28-ESR<3.2); Difference in Proportions = 26.3, 95% CI 2-sided [16.78 to 35.81] — Participants who took rescue therapy had the final value taken before rescue used for analysis at all ensuing time points

2. Secondary Outcome: Percentage of Participants Who Remained in Remission at Week 52 (DAS28-ESR)
Description: Proportion of participants who remained in Remission (DAS28-ESR <2.6) at Week 52.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
Percentage of participants | 53.2 | 29.5
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Test type: Superiority or Other; p = 0.019, Cochran-Mantel-Haenszel; The p-value from CMH test of general association was stratified by geographic region; Difference in proportions = 23.7, 95% CI 2-sided [6.83 to 40.61]

3. Secondary Outcome: Percentage of Participants Achieving LDA (DAS28-ESR and DAS28-C-reactive Protein [CRP]) at Each Visit During Period 1
Description: Proportion of participants who achieved LDA (DAS28-ESR and DAS28-CRP at each visit during period 1 is presented below.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: The FAS for Period 1 (Open Label FAS) included all randomized participants who had at least one dose of open label study drug during Period 1 (ie, ETN or MTX).
Measure: Number; unit: Percentage of participants
Groups:
- Open-Label Treatment: Participants in open-label treatment received ETN 50 mg QW with MTX (with or without other DMARDs).
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
Percentage of participants
  DAS28-ESR Week 4 (N= 473) | 9.5
  DAS28-CRP Week 4 (N= 465) | 20.6
  DAS28-ESR Week 8 (N= 473) | 20.3
  DAS28-CRP Week 8 (N= 471) | 34.6
  DAS28-ESR Week 16 (N= 473) | 32.8
  DAS28-CRP Week 16 (N= 472) | 52.8
  DAS28-ESR Week 24 (N= 473) | 72.1
  DAS28-CRP Week 24 (N= 472) | 72.5

4. Secondary Outcome: Percentage of Participants Achieving LDA (DAS28-ESR and DAS28-CRP) at Each Visit During Period 2
Description: Proportion of participants who achieved LDA (DAS28-ESR and DAS28-CRP at each visit during period 2 is presented below.
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
Percentage of participants
  DAS28-ESR Baseline (N= 163, 168) | 0.0 | 0.6
  DAS28-CRP Baseline (N= 163, 168) | 0.6 | 0.0
  DAS28-ESR Week 24 (N= 163, 168) | 100.0 | 100.0
  DAS28-CRP Week 24 (N= 163, 168) | 87.7 | 85.1
  DAS28-ESR Week 28 (N= 163, 168) | 62.6 | 41.1
  DAS28-CRP Week 28 (N= 160, 166) | 74.4 | 55.4
  DAS28-ESR Week 36 (N= 163, 168) | 55.2 | 24.4
  DAS28-CRP Week 36 (N= 162, 167) | 69.1 | 41.9
  DAS28-ESR Week 44 (N= 163, 168) | 51.5 | 20.2
  DAS28-CRP Week 44 (N= 162, 167) | 69.1 | 38.9
  DAS28-ESR Week 52 (N= 163, 168) | 43.6 | 17.3
  DAS28-CRP Week 52 (N= 162, 167) | 64.2 | 37.1
Statistical Analysis 1: Comparison: Etanercept vs Placebo; DAS28-ESR Baseline; Test type: Superiority or Other; p = 0.371, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = -0.6, 95% CI 2-sided [-1.76 to 0.57]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; DAS28-CRP Baseline; Test type: Superiority or Other; p = 0.358, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 0.6, 95% CI 2-sided [-0.59 to 1.81]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; DAS28-CRP Week 24; Test type: Superiority or Other; p = 0.667, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 2.6, 95% CI 2-sided [-4.76 to 9.98]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; DAS28-ESR Week 28; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 21.5, 95% CI 2-sided [10.99 to 32.02]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; DAS28-CRP Week 28; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 19.0, 95% CI 2-sided [8.81 to 29.10]
Statistical Analysis 6: Comparison: Etanercept vs Placebo; DAS28-ESR Week 36; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 30.8, 95% CI 2-sided [20.79 to 40.83]
Statistical Analysis 7: Comparison: Etanercept vs Placebo; DAS28-CRP Week 36; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 27.2, 95% CI 2-sided [16.89 to 37.54]
Statistical Analysis 8: Comparison: Etanercept vs Placebo; DAS28-ESR Week 44; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 31.3, 95% CI 2-sided [21.51 to 41.08]
Statistical Analysis 9: Comparison: Etanercept vs Placebo; DAS28-CRP Week 44; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 30.2, 95% CI 2-sided [19.95 to 40.47]
Statistical Analysis 10: Comparison: Etanercept vs Placebo; DAS28-ESR Week 52; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 26.3, 95% CI 2-sided [16.78 to 35.81]
Statistical Analysis 11: Comparison: Etanercept vs Placebo; DAS28-CRP Week 52; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 27.1, 95% CI 2-sided [16.67 to 37.47]

5. Secondary Outcome: Percentage of Participants Achieving Remission (DAS28-ESR and DAS28-CRP) at Each Visit During Period 1
Description: Proportion of participants who achieved remission (DAS28-ESR and DAS28-CRP at each visit during period 1 is presented below.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
Percentage of participants
  DAS28-ESR Week 4 (N= 473) | 4.0
  DAS28-CRP Week 4 (N= 465) | 9.0
  DAS28-ESR Week 8 (N= 473) | 8.9
  DAS28-CRP Week 8 (N= 471) | 17.8
  DAS28-ESR Week 16 (N= 473) | 13.5
  DAS28-CRP Week 16 (N= 472) | 31.1
  DAS28-ESR Week 24 (N= 473) | 26.6
  DAS28-CRP Week 24 (N= 472) | 49.8

6. Secondary Outcome: Percentage of Participants Achieving Remission (DAS28-ESR and DAS28-CRP) at Each Visit During Period 2
Description: Proportion of participants who achieved LDA (DAS28-ESR and DAS28-CRP at each visit during period 2 is presented below.
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
Percentage of participants
  DAS28-ESR Baseline (N= 163, 168) | 0.0 | 0.0
  DAS28-CRP Baseline (N= 163, 168) | 0.0 | 0.0
  DAS28-ESR Week 24 (N= 163, 168) | 38.0 | 36.3
  DAS28-CRP Week 24 (N= 163, 168) | 64.4 | 63.1
  DAS28-ESR Week 28 (N= 163, 168) | 32.5 | 20.2
  DAS28-CRP Week 28 (N= 160, 166) | 51.9 | 34.9
  DAS28-ESR Week 36 (N= 163, 168) | 31.9 | 17.3
  DAS28-CRP Week 36 (N= 162, 167) | 50.0 | 25.1
  DAS28-ESR Week 44 (N= 163, 168) | 30.7 | 11.9
  DAS28-CRP Week 44 (N= 162, 167) | 51.9 | 21.0
  DAS28-ESR Week 52 (N= 163, 168) | 33.7 | 13.1
  DAS28-CRP Week 52 (N= 162, 167) | 46.9 | 19.8
Statistical Analysis 1: Comparison: Etanercept vs Placebo; DAS28-CRP Week 24; Test type: Superiority or Other; p = 0.774, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 1.3, 95% CI 2-sided [-9.03 to 11.68]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; DAS28-ESR Week 28; Test type: Superiority or Other; p = 0.034, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 12.3, 95% CI 2-sided [2.86 to 21.69]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; DAS28-CRP Week 28; Test type: Superiority or Other; p = 0.020, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 16.9, 95% CI 2-sided [6.33 to 27.54]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; DAS28-ESR Week 36; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 14.6, 95% CI 2-sided [5.48 to 23.80]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; DAS28-CRP Week 36; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 24.9, 95% CI 2-sided [14.72 to 34.98]
Statistical Analysis 6: Comparison: Etanercept vs Placebo; DAS28-ESR Week 44; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 18.8, 95% CI 2-sided [10.16 to 27.38]
Statistical Analysis 7: Comparison: Etanercept vs Placebo; DAS28-CRP Week 44; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 30.9, 95% CI 2-sided [21.03 to 40.76]
Statistical Analysis 8: Comparison: Etanercept vs Placebo; DAS28-ESR Week 52; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 20.6, 95% CI 2-sided [11.78 to 29.52]
Statistical Analysis 9: Comparison: Etanercept vs Placebo; DAS28-CRP Week 52; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 27.2, 95% CI 2-sided [17.38 to 36.93]

7. Secondary Outcome: Change From Baseline in DAS28-CRP and DAS28-ESR in Period 1
Description: The DAS assessment is a derived measurement with differential weight given to each component. The DAS28-ESR and DAS28-CRP was calculated at every visit within the clinical database in period 1. The components of the DAS28 ESR score assessment are: Tender/ Painful Joint Count (28), Swollen Joint Count (28); ESR, Subject General Health VAS assessment. The components of the DAS28 CRP score assessment were: Tender/Painful Joint Count (28); Swollen Joint Count (28), hsCRP, and the Subject General Health VAS assessment. This efficacy measurement was made at every study visit.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
units on a scale
  DAS28-ESR Week 4 (N= 473) | -1.61 (1.08)
  DAS28-CRP Week 4 (N= 465) | -1.61 (1.05)
  DAS28-ESR Week 8 (N= 473) | -2.14 (1.18)
  DAS28-CRP Week 8 (N= 471) | -2.09 (1.14)
  DAS28-ESR Week 16 (N= 473) | -2.62 (1.26)
  DAS28-CRP Week 16 (N= 472) | -2.54 (1.21)
  DAS28-ESR Week 24 (N= 473) | -3.23 (1.35)
  DAS28-CRP Week 24 (N= 472) | -2.95 (1.27)

8. Secondary Outcome: Change From Baseline in DAS28-CRP and DAS28-ESR in Period 2
Description: The DAS assessment is a derived measurement with differential weight given to each component. The DAS28-ESR and DAS28-CRP was calculated at every visit within the clinical database in period 2. The components of the DAS28 ESR score assessment are: Tender/ Painful Joint Count (28), Swollen Joint Count (28); ESR, Subject General Health VAS assessment. The components of the DAS28 CRP score assessment were: Tender/Painful Joint Count (28); Swollen Joint Count (28), hsCRP, and the Subject General Health VAS assessment. This efficacy measurement was made at every study visit.
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
units on a scale
  DAS28-ESR Week 24 (N= 163, 168) | -3.79 (1.04) | -3.70 (0.99)
  DAS28-CRP Week 24 (N= 163, 168) | -3.36 (1.03) | -3.32 (1.05)
  DAS28-ESR Week 28 (N= 163, 168) | -3.35 (1.31) | -2.73 (1.43)
  DAS28-CRP Week 28 (N= 160, 166) | -3.06 (1.26) | -2.53 (1.40)
  DAS28-ESR Week 36 (N= 163, 168) | -3.20 (1.40) | -2.40 (1.49)
  DAS28-CRP Week 36 (N= 162, 167) | -2.97 (1.35) | -2.27 (1.48)
  DAS28-ESR Week 44 (N= 163, 168) | -3.15 (1.36) | -2.31 (1.49)
  DAS28-CRP Week 44 (N= 162, 167) | -2.95 (1.35) | -2.19 (1.50)
  DAS28-ESR Week 52 (N= 163, 168) | -3.08 (1.40) | -2.28 (1.46)
  DAS28-CRP Week 52 (N= 162, 167) | -2.92 (1.36) | -2.16 (1.45)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; DAS28-ESR Week 28; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-0.73 to -0.20]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; DAS28-CRP Week 28; Test type: Superiority or Other; p = 0.006, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.61 to -0.11]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; DAS28-ESR Week 36; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-0.96 to -0.39]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; DAS28-CRP Week 36; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-0.82 to -0.28]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; DAS28-ESR Week 44; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.03 to -0.46]
Statistical Analysis 6: Comparison: Etanercept vs Placebo; DAS28-CRP Week 44; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.65, 95% CI 2-sided [-0.92 to -0.37]
Statistical Analysis 7: Comparison: Etanercept vs Placebo; DAS28-ESR Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.69, 95% CI 2-sided [-0.98 to -0.40]
Statistical Analysis 8: Comparison: Etanercept vs Placebo; DAS28-CRP Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-0.91 to -0.36]

9. Secondary Outcome: Percentage of Participants Who Had a Recurrence of Disease Symptoms During Period 2, Based on the Protocol Criteria
Description: Flare is defined as the criteria of loss of LDA plus ≥0.6 unit worsening in DAS28-ESR score during period 2.
Time Frame: Baseline and Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
Percentage of participants | 52.1 | 79.8
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Test type: Superiority or Other; p < 0.001, Log Rank

10. Secondary Outcome: Percentage of Participants Achieving European League Against Rheumatism (EULAR) Good and or Moderate Responses (by Both DAS28-ESR and DAS28-CRP Scores) at Each Visit During Period 1.
Description: EULAR response is based on DAS28-ESR scores. The following good and moderate response is defined based on DAS28-ESR at endpoint (DAS28-ESR improvement at from Baseline in parenthesis): ≤3.2 units (>1.2 units) is good response; ≤3.2 units (0.6-1.2 units) are moderate response; ≤3.2 units (≤0.6 units) are no response.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
Percentage of participants
  Good Response: DAS28-ESR Week 4 (N= 473) | 9.5
  Good Response: DAS28-CRP Week 4 (N= 465) | 18.9
  Good Response: DAS28-ESR Week 8 (N= 473) | 19.5
  Good Response: DAS28-CRP Week 8 (N= 471) | 33.5
  Good Response: DAS28-ESR Week 16 (N= 473) | 32.3
  Good Response: DAS28-CRP Week 16 (N= 472) | 51.9
  Good Response: DAS28-ESR Week 24 (N= 473) | 71.5
  Good Response: DAS28-CRP Week 24 (N= 472) | 71.4
  Moderate Response: DAS28-ESR Week 4 (N= 473) | 69.1
  Moderate Response: DAS28-CRP Week 4 (N= 465) | 79.8
  Moderate Response: DAS28-ESR Week 8 (N= 473) | 86.9
  Moderate Response: DAS28-CRP Week 8 (N= 471) | 87.5
  Moderate Response: DAS28-ESR Week 16 (N= 473) | 92.0
  Moderate Response: DAS28-CRP Week 16 (N= 472) | 92.8
  Moderate Response: DAS28-ESR Week 24 (N= 473) | 94.1
  Moderate Response: DAS28-CRP Week 24 (N= 472) | 95.1

11. Secondary Outcome: Percentage of Participants Achieving EULAR Good and or Moderate Responses (by Both DAS28-ESR and DAS28-CRP Scores) at Each Visit During Period 2.
Description: as for outcome 10
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
Percentage of participants
  Good Response: DAS28-ESR Week 24 (N= 163, 168) | 99.4 | 99.4
  Good Response: DAS28-CRP Week 24 (N= 163, 168) | 86.5 | 85.1
  Good Response: DAS28-ESR Week 28 (N= 163, 168) | 62.6 | 41.1
  Good Response: DAS28-CRP Week 28 (N= 160, 166) | 73.1 | 54.8
  Good Response: DAS28-ESR Week 36 (N= 163, 168) | 55.2 | 23.8
  Good Response: DAS28-CRP Week 36 (N= 162, 167) | 67.9 | 40.7
  Good Response: DAS28-ESR Week 44 (N= 163, 168) | 50.9 | 19.6
  Good Response: DAS28-CRP Week 44 (N= 162, 167) | 68.5 | 37.7
  Good Response: DAS28-ESR Week 52 (N= 163, 168) | 42.9 | 16.7
  Good Response: DAS28-CRP Week 52 (N= 162, 167) | 63.0 | 35.9
  Moderate Response: DAS28-ESR Week 24 (N= 163, 168) | 100.0 | 100.0
  Moderate Response: DAS28-CRP Week 24 (N= 163, 168) | 100.0 | 100.0
  Moderate Response: DAS28-ESR Week 28 (N= 163, 168) | 95.7 | 87.5
  Moderate Response: DAS28-CRP Week 28 (N= 160, 166) | 96.9 | 90.4
  Moderate Response: DAS28-ESR Week 36 (N= 163, 168) | 93.9 | 83.9
  Moderate Response: DAS28-CRP Week 36 (N= 162, 167) | 94.4 | 85.6
  Moderate Response: DAS28-ESR Week 44 (N= 163, 168) | 93.3 | 81.5
  Moderate Response: DAS28-CRP Week 44 (N= 162, 167) | 95.1 | 84.4
  Moderate Response: DAS28-ESR Week 52 (N= 163, 168) | 93.3 | 82.1
  Moderate Response: DAS28-CRP Week 52 (N= 162, 167) | 95.7 | 84.4
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Good Response: DAS28-CRP Week 24; Test type: Superiority or Other; p = 0.961, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 1.4, 95% CI 2-sided [-6.13 to 8.90]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Good Response: DAS28-ESR Week 28; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 21.5, 95% CI 2-sided [10.99 to 32.02]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Good Response: DAS28-CRP Week 28; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 18.3, 95% CI 2-sided [8.08 to 28.53]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Good Response: DAS28-ESR Week 36; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 31.4, 95% CI 2-sided [21.42 to 41.39]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; Good Response: DAS28-CRP Week 36; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 27.2, 95% CI 2-sided [16.83 to 37.54]
Statistical Analysis 6: Comparison: Etanercept vs Placebo; Good Response: DAS28-ESR Week 44; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 31.3, 95% CI 2-sided [21.53 to 41.02]
Statistical Analysis 7: Comparison: Etanercept vs Placebo; Good Response: DAS28-CRP Week 44; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 30.8, 95% CI 2-sided [20.54 to 41.05]
Statistical Analysis 8: Comparison: Etanercept vs Placebo; Good Response: DAS28-ESR Week 52; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 26.3, 95% CI 2-sided [16.82 to 35.74]
Statistical Analysis 9: Comparison: Etanercept vs Placebo; Good Response: DAS28-CRP Week 52; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 27.0, 95% CI 2-sided [16.63 to 37.44]
Statistical Analysis 10: Comparison: Etanercept vs Placebo; Good Response: DAS28-ESR Week 24; Test type: Superiority or Other; p = 0.766, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in Proportions = -0.0, 95% CI 2-sided [-1.69 to 1.65]
Statistical Analysis 11: Comparison: Etanercept vs Placebo; Moderate Response: DAS28-ESR Week 28; Test type: Superiority or Other; p = 0.091, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in Proportions = 8.2, 95% CI 2-sided [2.32 to 14.10]
Statistical Analysis 12: Comparison: Etanercept vs Placebo; Moderate Response: DAS28-CRP Week 28; Test type: Superiority or Other; p = 0.227, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 6.5, 95% CI 2-sided [1.28 to 11.75]
Statistical Analysis 13: Comparison: Etanercept vs Placebo; Moderate Response: DAS28-ESR Week 36; Test type: Superiority or Other; p = 0.072, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 9.9, 95% CI 2-sided [3.27 to 16.60]
Statistical Analysis 14: Comparison: Etanercept vs Placebo; Moderate Response: DAS28-CRP Week 36; Test type: Superiority or Other; p = 0.108, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 8.8, 95% CI 2-sided [2.43 to 15.20]
Statistical Analysis 15: Comparison: Etanercept vs Placebo; Moderate Response: DAS28-ESR Week 44; Test type: Superiority or Other; p = 0.035, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 11.7, 95% CI 2-sided [4.69 to 18.72]
Statistical Analysis 16: Comparison: Etanercept vs Placebo; Moderate Response: DAS28-ESR Week 44; Test type: Superiority or Other; p = 0.030, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 10.6, 95% CI 2-sided [4.20 to 17.06]
Statistical Analysis 17: Comparison: Etanercept vs Placebo; Moderate Response: DAS28-ESR Week 52; Test type: Superiority or Other; p = 0.048, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 11.1, 95% CI 2-sided [4.15 to 18.06]
Statistical Analysis 18: Comparison: Etanercept vs Placebo; Moderate Response: DAS28-CRP Week 52; Test type: Superiority or Other; p = 0.016, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 11.2, 95% CI 2-sided [4.92 to 17.58]

12. Secondary Outcome: Percentage of Participants Achieving LDA or Remission Based on Clinical Disease Activity Index (CDAI) and Simplified Disease Activity Index (SDAI) at Each Visit During Period 1.
Description: SDAI and CDAI are defined as:
  1) SDAI = DAS28 prorated Swollen Joint Count (0-28) + DAS28 prorated Tender Joint Count (0-28) + Physician Global Assessment of arthritis (0-10) + Subject Global Assessment of arthritis (0-10) + hs CRP (in mg/dL) in Period 1. 2) CDAI = DAS28 prorated Swollen Joint Count (0-28) + DAS28 prorated Tender Joint Count (0 28) + Physician Global Assessment of arthritis (0-10) + Subject Global Assessment of arthritis (0-10) in Period 1.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
Percentage of participants
  CDAI: LDA Baseline (N= 478) | 0.4
  CDAI: LDA Week 4 (N= 473) | 16.7
  CDAI: LDA Week 8 (N= 473) | 33.8
  CDAI: LDA Week 16 (N= 473) | 53.9
  CDAI: LDA Week 24 (N= 473) | 75.7
  CDAI: Remission: Baseline (N= 478) | 0.0
  CDAI: Remission: Week 4 (N= 473) | 0.4
  CDAI: Remission: Week 8 (N= 473) | 1.7
  CDAI: Remission: Week 16 (N= 473) | 6.1
  CDAI: Remission: Week 24 (N= 473) | 10.8
  SDAI: LDA: Baseline (N= 478) | 0.2
  SDAI: LDA: Week 4 (N= 465) | 16.1
  SDAI: LDA: Week 8 (N= 471) | 32.5
  SDAI: LDA: Week 16 (N= 472) | 52.3
  SDAI: LDA: Week 24 (N= 472) | 72.5
  SDAI: Remission: Baseline (N= 478) | 0.0
  SDAI: Remission: Week 4 (N= 465) | 0.6
  SDAI: Remission: Week 8 (N= 471) | 1.9
  SDAI: Remission: Week 16 (N= 472) | 6.8
  SDAI: Remission: Week 24 (N= 472) | 14.0

13. Secondary Outcome: Percentage of Participants Achieving LDA or Remission Based on CDAI and SDAI at Each Visit During Period 2.
Description: SDAI and CDAI are defined as:
  1) SDAI = DAS28 prorated Swollen Joint Count (0-28) + DAS28 prorated Tender Joint Count (0-28) + Physician Global Assessment of arthritis (0-10) + Subject Global Assessment of arthritis (0-10) + hs CRP (in mg/dL) in Period 2. 2) CDAI = DAS28 prorated Swollen Joint Count (0-28) + DAS28 prorated Tender Joint Count (0 28) + Physician Global Assessment of arthritis (0-10) + Subject Global Assessment of arthritis (0-10) in Period 2.
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
Percentage of participants
  CDAI: LDA Baseline (N= 163, 168) | 0.6 | 0.0
  CDAI: LDA Week 24 (N= 163, 168) | 93.9 | 90.5
  CDAI: LDA Week 28 (N= 163, 168) | 76.1 | 57.7
  CDAI: LDA Week 36 (N= 163, 168) | 71.2 | 47.0
  CDAI: LDA Week 44 (N= 163, 168) | 70.6 | 43.5
  CDAI: LDA Week 52 (N= 163, 168) | 66.9 | 42.9
  CDAI: Remission: Baseline (N= 163, 168) | 0.0 | 0.0
  CDAI: Remission: Week 24 (N= 163, 168) | 16.6 | 14.3
  CDAI: Remission: Week 28 (N= 163, 168) | 14.7 | 14.3
  CDAI: Remission: Week 36 (N= 163, 168) | 20.9 | 12.5
  CDAI: Remission: Week 44 (N= 163, 168) | 22.1 | 12.5
  CDAI: Remission: Week 52 (N= 163, 168) | 20.9 | 11.9
  SDAI: LDA: Baseline (N= 163, 168) | 0.6 | 0.0
  SDAI: LDA: Week 24 (N= 163, 168) | 90.2 | 86.9
  SDAI: LDA: Week 28 (N= 160, 166) | 73.1 | 55.4
  SDAI: LDA: Week 36 (N= 162, 167) | 69.8 | 42.5
  SDAI: LDA: Week 44 (N= 162, 167) | 69.8 | 42.5
  SDAI: LDA: Week 52 (N= 162, 167) | 69.8 | 37.7
  SDAI: Remission: Baseline (N= 163, 168) | 0.0 | 0.0
  SDAI: Remission: Week 24 (N= 163, 168) | 20.9 | 17.9
  SDAI: Remission: Week 28 (N= 160, 166) | 16.3 | 16.3
  SDAI: Remission: Week 36 (N= 162, 167) | 22.8 | 12.6
  SDAI: Remission: Week 44 (N= 162, 167) | 22.2 | 13.2
  SDAI: Remission: Week 52 (N= 162, 167) | 25.3 | 13.2
Statistical Analysis 1: Comparison: Etanercept vs Placebo; CDAI: LDA Baseline; Test type: Superiority or Other; p = 0.358, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 0.6, 95% CI 2-sided [-0.59 to 1.81]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; CDAI: LDA: Week 24; Test type: Superiority or Other; p = 0.341, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 3.4, 95% CI 2-sided [-2.38 to 9.16]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; CDAI: LDA: Week 28; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 18.3, 95% CI 2-sided [8.40 to 28.27]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; CDAI: LDA: Week 36; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 24.1, 95% CI 2-sided [13.88 to 34.40]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; CDAI: LDA: Week 44; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 27.1, 95% CI 2-sided [16.85 to 37.35]
Statistical Analysis 6: Comparison: Etanercept vs Placebo; CDAI: LDA: Week 52; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 24.0, 95% CI 2-sided [13.61 to 34.42]
Statistical Analysis 7: Comparison: Etanercept vs Placebo; CDAI: Remission: Week 24; Test type: Superiority or Other; p = 0.774, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 2.3, 95% CI 2-sided [-5.50 to 10.06]
Statistical Analysis 8: Comparison: Etanercept vs Placebo; CDAI: Remission: Week 28; Test type: Superiority or Other; p = 0.645, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 0.4, 95% CI 2-sided [-7.15 to 8.03]
Statistical Analysis 9: Comparison: Etanercept vs Placebo; CDAI: Remission: Week 36; Test type: Superiority or Other; p = 0.080, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 8.4, 95% CI 2-sided [0.36 to 16.35]
Statistical Analysis 10: Comparison: Etanercept vs Placebo; CDAI: Remission: Week 44; Test type: Superiority or Other; p = 0.025, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 9.6, 95% CI 2-sided [1.49 to 17.68]
Statistical Analysis 11: Comparison: Etanercept vs Placebo; CDAI: Remission: Week 52; Test type: Superiority or Other; p = 0.088, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 9.0, 95% CI 2-sided [1.02 to 16.88]
Statistical Analysis 12: Comparison: Etanercept vs Placebo; SDAI: LDA: Baseline; Test type: Superiority or Other; p = 0.358, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 0.6, 95% CI 2-sided [-0.59 to 1.81]
Statistical Analysis 13: Comparison: Etanercept vs Placebo; SDAI: LDA: Week 24; Test type: Superiority or Other; p = 0.258, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 3.3, 95% CI 2-sided [-3.57 to 10.13]
Statistical Analysis 14: Comparison: Etanercept vs Placebo; SDAI: LDA: Week 28; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 17.7, 95% CI 2-sided [7.49 to 27.92]
Statistical Analysis 15: Comparison: Etanercept vs Placebo; SDAI: LDA: Week 36; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 27.2, 95% CI 2-sided [16.93 to 37.55]
Statistical Analysis 16: Comparison: Etanercept vs Placebo; SDAI: LDA: Week 44; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 32.0, 95% CI 2-sided [21.83 to 42.23]
Statistical Analysis 17: Comparison: Etanercept vs Placebo; SDAI: LDA: Week 52; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 28.3, 95% CI 2-sided [18.00 to 38.69]
Statistical Analysis 18: Comparison: Etanercept vs Placebo; SDAI: Remission: Week 24; Test type: Superiority or Other; p = 0.672, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 3.0, 95% CI 2-sided [-5.51 to 11.51]
Statistical Analysis 19: Comparison: Etanercept vs Placebo; SDAI: Remission: Week 28; Test type: Superiority or Other; p = 0.556, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = -0.0, 95% CI 2-sided [-8.03 to 8.00]
Statistical Analysis 20: Comparison: Etanercept vs Placebo; SDAI: Remission: Week 36; Test type: Superiority or Other; p = 0.022, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 10.3, 95% CI 2-sided [2.07 to 18.45]
Statistical Analysis 21: Comparison: Etanercept vs Placebo; SDAI: Remission: Week 44; Test type: Superiority or Other; p = 0.047, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 9.0, 95% CI 2-sided [0.85 to 17.25]
Statistical Analysis 22: Comparison: Etanercept vs Placebo; SDAI: Remission: Week 52; Test type: Superiority or Other; p = 0.031, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 12.1, 95% CI 2-sided [3.70 to 20.57]

14. Secondary Outcome: Change of CDAI and SDAI at Each Visit During Period 1.
Description: as for outcome 12
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
units on a scale
  CDAI Week 4 (N= 473) | -16.78 (11.72)
  CDAI Week 8 (N= 473) | -21.69 (12.40)
  CDAI Week 16 (N= 473) | -25.77 (13.19)
  CDAI Week 24 (N= 473) | -29.25 (13.66)
  SDAI Week 4 (N= 465) | -18.19 (12.44)
  SDAI Week 8 (N= 471) | -23.06 (12.89)
  SDAI Week 16 (N= 472) | -27.17 (13.61)
  SDAI Week 24 (N= 472) | -30.56 (14.27)

15. Secondary Outcome: Change of CDAI and SDAI at Each Visit During Period 2
Description: as for outcome 13
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
units on a scale
  CDAI: Week 24 (N= 163, 168) | -32.11 (12.06) | -32.23 (12.49)
  CDAI: Week 28 (N= 163, 168) | -29.62 (13.10) | -26.49 (15.87)
  CDAI: Week 36 (N= 163, 168) | -28.71 (13.56) | -24.33 (16.45)
  CDAI: Week 44 (N= 163, 168) | -28.63 (13.58) | -23.81 (16.48)
  CDAI: Week 52 (N= 163, 168) | -28.30 (13.61) | -23.52 (15.98)
  SDAI: Week 24 (N= 163, 168) | -33.61 (12.07) | -33.68 (13.03)
  SDAI: Week 28 (N= 160, 166) | -31.07 (13.58) | -27.58 (16.50)
  SDAI: Week 36 (N= 162, 167) | -30.20 (14.05) | -25.44 (17.17)
  SDAI: Week 44 (N= 162, 167) | -30.21 (14.14) | -24.85 (17.29)
  SDAI: Week 52 (N= 162, 167) | -29.86 (14.03) | -24.57 (16.79)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; CDAI: Week 28; Test type: Superiority or Other; p = 0.049, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.10, 95% CI 2-sided [-4.19 to -0.01]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; CDAI: Week 36; Test type: Superiority or Other; p = 0.005, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.38, 95% CI 2-sided [-5.72 to -1.05]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; CDAI: Week 44; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.02, 95% CI 2-sided [-6.37 to -1.67]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; CDAI: Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.02, 95% CI 2-sided [-6.36 to -1.68]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; SDAI: Week 28; Test type: Superiority or Other; p = 0.047, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.22, 95% CI 2-sided [-4.40 to -0.03]
Statistical Analysis 6: Comparison: Etanercept vs Placebo; SDAI: Week 36; Test type: Superiority or Other; p = 0.004, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.54, 95% CI 2-sided [-5.97 to -1.12]
Statistical Analysis 7: Comparison: Etanercept vs Placebo; SDAI: Week 44; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.33, 95% CI 2-sided [-6.78 to -1.88]
Statistical Analysis 8: Comparison: Etanercept vs Placebo; SDAI: Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.27, 95% CI 2-sided [-6.70 to -1.84]

16. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) ACR20, ACR50, ACR70 and ACR90 (by 66/68 Joint Counts) During Period 1 at Each Visit.
Description: A 66 swollen and 68 tender joint count was used for calculating ACR responses. The ACR's definition for calculating improvement in RA (ACR20) was calculated as a 20% improvement in tender and swollen joint counts and 20% improvement in 3 of the 5 remaining ACR core set measures: subject and physician global assessments of arthritis, pain, disability, and an acute phase reactant. Similarly, ACR50, ACR70 and ACR90 were calculated with the respective percent improvement. This efficacy measurement was made at every study visit.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
percentage of participants
  ACR 20: Week 4 (N= 469) | 58.6 (1.08)
  ACR 20: Week 8 (N= 469) | 73.1 (1.05)
  ACR 20: Week 16 (N= 469) | 83.6 (1.18)
  ACR 20: Week 24 (N= 469) | 87.8 (1.14)
  ACR 50: Week 4 (N= 469) | 19.8 (1.26)
  ACR 50: Week 8 (N= 469) | 35.8 (1.21)
  ACR 50: Week 16 (N= 469) | 55.2 (1.35)
  ACR 50: Week 24 (N= 469) | 72.5 (1.27)
  ACR 70: Week 4 (N= 469) | 4.3
  ACR 70: Week 8 (N= 469) | 11.1
  ACR 70: Week 16 (N= 469) | 23.7
  ACR 70: Week 24 (N= 469) | 39.4
  ACR 90: Week 4 (N= 469) | 0.0
  ACR 90: Week 8 (N= 469) | 0.4
  ACR 90: Week 16 (N= 469) | 1.5
  ACR 90: Week 24 (N= 469) | 5.8

17. Secondary Outcome: Percentage of Participants Achieving ACR20, ACR50, ACR70 and ACR90 (by 66/68 Joint Counts) During Period 2 at Each Visit.
Description: as for outcome 16
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
Percentage of participants
  ACR 20: Week 24 (N= 161, 168) | 96.3 | 96.4
  ACR 20: Week 28 (N= 161, 168) | 91.3 | 81.5
  ACR 20: Week 36 (N= 161, 168) | 88.2 | 76.8
  ACR 20: Week 44 (N= 161, 168) | 86.3 | 76.2
  ACR 20: Week 52 (N= 161, 168) | 87.0 | 76.2
  ACR 50: Week 24 (N= 161, 168) | 88.2 | 85.7
  ACR 50: Week 28 (N= 161, 168) | 75.2 | 63.7
  ACR 50: Week 36 (N= 161, 168) | 68.9 | 51.8
  ACR 50: Week 44 (N= 161, 168) | 69.6 | 50.6
  ACR 50: Week 52 (N= 161, 168) | 68.3 | 50.6
  ACR 70: Week 24 (N= 161, 168) | 49.7 | 52.4
  ACR 70: Week 28 (N= 161, 168) | 41.0 | 33.9
  ACR 70: Week 36 (N= 161, 168) | 44.7 | 27.4
  ACR 70: Week 44 (N= 161, 168) | 43.5 | 25.0
  ACR 70: Week 52 (N= 161, 168) | 41.0 | 25.0
  ACR 90: Week 24 (N= 161, 168) | 8.1 | 8.3
  ACR 90: Week 28 (N= 161, 168) | 8.7 | 5.4
  ACR 90: Week 36 (N= 161, 168) | 11.8 | 5.4
  ACR 90: Week 44 (N= 161, 168) | 9.3 | 4.8
  ACR 90: Week 52 (N= 161, 168) | 13.0 | 7.1
Statistical Analysis 1: Comparison: Etanercept vs Placebo; ACR 20: Week 24; Test type: Superiority or Other; p = 0.742, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = -0.2, 95% CI 2-sided [-4.21 to 3.90]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; ACR 20: Week 28; Test type: Superiority or Other; p = 0.143, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 9.8, 95% CI 2-sided [2.45 to 17.06]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; ACR 20: Week 36; Test type: Superiority or Other; p = 0.111, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 11.4, 95% CI 2-sided [3.31 to 19.51]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; ACR 20: Week 44; Test type: Superiority or Other; p = 0.175, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 10.1, 95% CI 2-sided [1.80 to 18.49]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; ACR 20: Week 52; Test type: Superiority or Other; p = 0.088, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 10.8, 95% CI 2-sided [2.49 to 19.05]
Statistical Analysis 6: Comparison: Etanercept vs Placebo; ACR 50: Week 24; Test type: Superiority or Other; p = 0.584, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 2.5, 95% CI 2-sided [-4.78 to 9.75]
Statistical Analysis 7: Comparison: Etanercept vs Placebo; ACR 50: Week 28; Test type: Superiority or Other; p = 0.226, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 11.5, 95% CI 2-sided [1.59 to 21.34]
Statistical Analysis 8: Comparison: Etanercept vs Placebo; ACR 50: Week 36; Test type: Superiority or Other; p = 0.012, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 17.2, 95% CI 2-sided [6.76 to 27.56]
Statistical Analysis 9: Comparison: Etanercept vs Placebo; ACR 50: Week 44; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 19.0, 95% CI 2-sided [8.59 to 29.35]
Statistical Analysis 10: Comparison: Etanercept vs Placebo; ACR 50: Week 52; Test type: Superiority or Other; p = 0.014, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in Proportions = 17.7, 95% CI 2-sided [7.30 to 28.16]
Statistical Analysis 11: Comparison: Etanercept vs Placebo; ACR 70: Week 24; Test type: Superiority or Other; p = 0.702, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in Proportions = -2.7, 95% CI 2-sided [-13.49 to 8.11]
Statistical Analysis 12: Comparison: Etanercept vs Placebo; ACR 70: Week 28; Test type: Superiority or Other; p = 0.378, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 7.1, 95% CI 2-sided [-3.37 to 17.50]
Statistical Analysis 13: Comparison: Etanercept vs Placebo; ACR 70: Week 36; Test type: Superiority or Other; p = 0.004, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 17.3, 95% CI 2-sided [7.12 to 27.56]
Statistical Analysis 14: Comparison: Etanercept vs Placebo; ACR 70: Week 44; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 18.5, 95% CI 2-sided [8.40 to 28.55]
Statistical Analysis 15: Comparison: Etanercept vs Placebo; ACR 70: Week 52; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 16.0, 95% CI 2-sided [5.96 to 26.02]
Statistical Analysis 16: Comparison: Etanercept vs Placebo; ACR 90: Week 24; Test type: Superiority or Other; p = 0.921, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = -0.3, 95% CI 2-sided [-6.19 to 5.67]
Statistical Analysis 17: Comparison: Etanercept vs Placebo; ACR 90: Week 28; Test type: Superiority or Other; p = 0.410, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 3.3, 95% CI 2-sided [-2.19 to 8.86]
Statistical Analysis 18: Comparison: Etanercept vs Placebo; ACR 90: Week 36; Test type: Superiority or Other; p = 0.073, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 6.4, 95% CI 2-sided [0.41 to 12.48]
Statistical Analysis 19: Comparison: Etanercept vs Placebo; ACR 90: Week 44; Test type: Superiority or Other; p = 0.219, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 4.6, 95% CI 2-sided [-0.97 to 10.08]
Statistical Analysis 20: Comparison: Etanercept vs Placebo; ACR 90: Week 52; Test type: Superiority or Other; p = 0.196, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in proportions = 5.9, 95% CI 2-sided [-0.60 to 12.40]

18. Secondary Outcome: Change in the Tender and Swollen Joint Counts at Each Visit During Period 1 (Using 28 Joint Count as Well as 66/68 Joint Counts).
Description: A total of 66 swollen and 68 tender joints were assessed for tenderness/pain and swelling by the same qualified personnel (when possible) at each visit. For ACR responses, a 66/68 joint count was used. For DAS28-ESR, Simplified Disease Activity Index (SDAI), and Clinical Disease Activity Index (CDAI) calculations, the 28 joint count was used, which included: shoulders, elbows, wrists, metacarpophalangeal (MCP) joints, proximal interphalangeal (PIP) joints, and knees.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
Units on a scale
  28 Tender Joint Count: Week 4 | -6.49 (6.07)
  28 Tender Joint Count: Week 8 | -8.59 (6.32)
  28 Tender Joint Count: Week 16 | -10.12 (6.82)
  28 Tender Joint Count: Week 24 | -11.50 (6.79)
  28 Swollen Joint Count: Week 4 | -5.52 (5.02)
  28 Swollen Joint Count: Week 8 | -7.04 (5.36)
  28 Swollen Joint Count: Week 16 | -8.21 (5.44)
  28 Swollen Joint Count: Week 24 | -9.01 (5.65)
  68 Tender Joint Count: Week 4 | -9.71 (10.00)
  68 Tender Joint Count: Week 8 | -13.02 (10.95)
  68 Tender Joint Count: Week 16 | -15.21 (11.90)
  68 Tender Joint Count: Week 24 | -17.41 (12.72)
  68 Swollen Joint Count: Week 4 | -7.12 (6.86)
  68 Swollen Joint Count: Week 8 | -9.03 (7.54)
  68 Swollen Joint Count: Week 16 | -10.49 (7.62)
  68 Swollen Joint Count: Week 24 | -11.53 (8.65)

19. Secondary Outcome: Change in the Tender and Swollen Joint Counts at Each Visit During Period 2 (Using 28 Joint Count as Well as 66/68 Joint Counts).
Description: as for outcome 18
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
units on a scale
  28 Tender Joint Count: Week 24 | -12.65 (6.25) | -12.35 (6.45)
  28 Tender Joint Count: Week 28 | -11.69 (6.74) | -10.08 (7.84)
  28 Tender Joint Count: Week 36 | -11.22 (6.91) | -9.23 (8.07)
  28 Tender Joint Count: Week 44 | -11.19 (6.82) | -8.97 (8.01)
  28 Tender Joint Count: Week 52 | -11.03 (6.81) | -8.78 (7.83)
  28 Swollen Joint Count: Week 24 | -9.78 (5.16) | -9.98 (5.58)
  28 Swollen Joint Count: Week 28 | -8.97 (5.27) | -8.70 (5.94)
  28 Swollen Joint Count: Week 36 | -8.64 (5.51) | -8.16 (6.04)
  28 Swollen Joint Count: Week 44 | -8.71 (5.52) | -8.03 (6.08)
  28 Swollen Joint Count: Week 52 | -8.59 (5.42) | -7.98 (6.05)
  68 Tender Joint Count: Week 24 | -18.31 (12.13) | -18.19 (12.03)
  68 Tender Joint Count: Week 28 | -17.02 (12.48) | -15.20 (13.95)
  68 Tender Joint Count: Week 36 | -17.27 (12.55) | -17.13 (14.28)
  68 Tender Joint Count: Week 44 | -18.67 (12.90) | -18.82 (14.71)
  68 Tender Joint Count: Week 52 | -17.88 (13.21) | -17.61 (12.57)
  68 Swollen Joint Count: Week 24 | -12.09 (7.76) | -12.40 (8.45)
  68 Swollen Joint Count: Week 28 | -11.23 (7.77) | -10.81 (8.66)
  68 Swollen Joint Count: Week 36 | -11.26 (8.05) | -10.67 (8.59)
  68 Swollen Joint Count: Week 44 | -12.00 (8.03) | -11.63 (8.58)
  68 Swollen Joint Count: Week 52 | -11.98 (8.17) | -11.89 (8.91)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; 28 Tender Joint Count: Week 28; Test type: Superiority or Other; p = 0.062, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.90, 95% CI 2-sided [-1.84 to 0.05]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; 28 Tender Joint Count: Week 36; Test type: Superiority or Other; p = 0.015, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.34, 95% CI 2-sided [-2.41 to -0.27]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; 28 Tender Joint Count: Week 44; Test type: Superiority or Other; p = 0.003, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.65, 95% CI 2-sided [-2.72 to -0.57]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; 28 Tender Joint Count: Week 52; Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.75, 95% CI 2-sided [-2.85 to -0.66]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; 28 Swollen Joint Count: Week 28; Test type: Superiority or Other; p = 0.680, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.77 to 0.50]
Statistical Analysis 6: Comparison: Etanercept vs Placebo; 28 Swollen Joint Count: Week 36; Test type: Superiority or Other; p = 0.437, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.29, 95% CI 2-sided [-1.04 to 0.45]
Statistical Analysis 7: Comparison: Etanercept vs Placebo; 28 Swollen Joint Count: Week 44; Test type: Superiority or Other; p = 0.131, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.31 to 0.17]
Statistical Analysis 8: Comparison: Etanercept vs Placebo; 28 Swollen Joint Count: Week 52; Test type: Superiority or Other; p = 0.199, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-1.22 to 0.25]
Statistical Analysis 9: Comparison: Etanercept vs Placebo; 68 Tender Joint Count: Week 28; Test type: Superiority or Other; p = 0.115, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.16, 95% CI 2-sided [-2.60 to 0.28]
Statistical Analysis 10: Comparison: Etanercept vs Placebo; 68 Tender Joint Count: Week 36; Test type: Superiority or Other; p = 0.017, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.88, 95% CI 2-sided [-3.42 to -0.35]
Statistical Analysis 11: Comparison: Etanercept vs Placebo; 68 Tender Joint Count: Week 44; Test type: Superiority or Other; p = 0.004, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.34, 95% CI 2-sided [-3.91 to -0.76]
Statistical Analysis 12: Comparison: Etanercept vs Placebo; 68 Tender Joint Count: Week 52; Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.58, 95% CI 2-sided [-4.19 to -0.97]
Statistical Analysis 13: Comparison: Etanercept vs Placebo; 68 Swollen Joint Count: Week 28; Test type: Superiority or Other; p = 0.368, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-1.13 to 0.42]
Statistical Analysis 14: Comparison: Etanercept vs Placebo; 68 Swollen Joint Count: Week 36; Test type: Superiority or Other; p = 0.208, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-1.46 to 0.32]
Statistical Analysis 15: Comparison: Etanercept vs Placebo; 68 Swollen Joint Count: Week 44; Test type: Superiority or Other; p = 0.064, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.84, 95% CI 2-sided [-1.73 to 0.05]
Statistical Analysis 16: Comparison: Etanercept vs Placebo; 68 Swollen Joint Count: Week 52; Test type: Superiority or Other; p = 0.081, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.66 to 0.10]

20. Secondary Outcome: Change in the Physician Global Assessment of Arthritis at Each Visit During Period 1
Description: The investigator estimated the subject's overall disease activity over the last 2 to 3 days (independent of the Subject Global Assessment of arthritis) using a scale between 0 (no disease activity) and 10 (extreme disease activity) and marking one number with an 'X'.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
units on a scale
  Week 4 (N= 473) | -2.60 (1.78)
  Week 8 (N= 473) | -3.46 (1.90)
  Week 16 (N= 473) | -4.12 (1.96)
  Week 24 (N= 473) | -4.79 (2.02)

21. Secondary Outcome: Change in the Physician Global Assessment of Arthritis at Each Visit During Period 2
Description: as for outcome 20
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
units on a scale
  Week 24 | -5.28 (1.56) | -5.26 (1.78)
  Week 28 | -4.93 (1.78) | -4.23 (2.43)
  Week 36 | -4.83 (1.86) | -3.89 (2.48)
  Week 44 | -4.82 (2.02) | -3.79 (2.53)
  Week 52 | -4.77 (2.03) | -3.74 (2.43)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 28; Test type: Superiority or Other; p = 0.005, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.53, 95% CI 2-sided [-0.90 to -0.16]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 36; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.78, 95% CI 2-sided [-1.18 to -0.38]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Week 44; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.94, 95% CI 2-sided [-1.35 to -0.54]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-1.33 to -0.53]

22. Secondary Outcome: Change in the Subject Global Assessment of Arthritis in Period 1
Description: Subjects assessed their overall disease activity over the last 2 to 3 days using a scale between 0 (no disease activity) and 10 (extreme disease activity), which corresponded to the magnitude of their pain) and marked one number with an 'X'.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
units on a scale
  Week 4 (N= 473) | -2.18 (2.21)
  Week 8 (N= 473) | -2.60 (2.34)
  Week 16 (N= 473) | -3.32 (2.44)
  Week 24 (N= 473) | -3.97 (2.60)

23. Secondary Outcome: Change in the Subject Global Assessment of Arthritis in Period 2
Description: as for outcome 22
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
units on a scale
  Week 24 | -4.39 (2.43) | -4.64 (2.16)
  Week 28 | -4.03 (2.70) | -3.48 (2.94)
  Week 36 | -4.02 (2.71) | -3.05 (2.94)
  Week 44 | -3.92 (2.79) | -3.02 (2.91)
  Week 52 | -3.91 (2.84) | -3.02 (2.91)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 28; Test type: Superiority or Other; p = 0.048, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.50, 95% CI 2-sided [-1.00 to -0.01]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 36; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.93, 95% CI 2-sided [-1.44 to -0.43]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Week 44; Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-1.33 to -0.33]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Week 52; Test type: Superiority or Other; p = 0.002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.82, 95% CI 2-sided [-1.33 to -0.31]

24. Secondary Outcome: Change in Morning Stiffness (Measured in Minutes) at Each Visit During Period 1
Description: Morning stiffness was defined as stiffness in and around the joints, lasting at least 1 hour before maximal improvement. Participants assessed their overall disease activity over the last 2 to 3 days using a scale between 0 (no disease activity) and 10 (extreme disease activity), which corresponded to the magnitude of their pain) and marked one number with an 'X'.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
minutes
  Week 4 (N= 467) | -78.56 (143.68)
  Week 8 (N= 467) | -90.58 (147.42)
  Week 16 (N= 467) | -102.25 (158.76)
  Week 24 (N= 467) | -109.32 (183.15)

25. Secondary Outcome: Change in Morning Stiffness (Measured in Minutes) at Each Visit During Period 2
Description: as for outcome 24
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
minutes
  Week 24 (N= 163, 166) | -118.30 (171.15) | -121.93 (186.17)
  Week 28 (N= 163, 166) | -134.42 (224.70) | -109.57 (163.79)
  Week 36 (N= 163, 166) | -132.05 (224.86) | -104.40 (164.13)
  Week 44 (N= 163, 166) | -129.86 (223.78) | -103.14 (162.65)
  Week 52 (N= 163, 166) | -129.49 (223.68) | -100.31 (153.62)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 28; Test type: Superiority or Other; p = 0.033, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -14.11, 95% CI 2-sided [-27.07 to -1.16]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 36; Test type: Superiority or Other; p = 0.013, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -17.04, 95% CI 2-sided [-30.39 to -3.68]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Week 44; Test type: Superiority or Other; p = 0.019, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -16.54, 95% CI 2-sided [-30.35 to -2.73]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Week 52; Test type: Superiority or Other; p = 0.007, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -19.66, 95% CI 2-sided [-33.78 to -5.54]

26. Secondary Outcome: Change in the Subject General Health Visual Analog Scale (VAS) and Pain VAS at Each Visit During Period 1
Description: Participants were asked to answer the question "In general how would you rate your health over the last 2 3 weeks?" by marking a vertical line at the appropriate position through the 100 mm VAS. The length on the line was measured from the left (in mm). For Pain VAS, participants assessed the severity of their arthritis pain during the last 2 to 3 days using a 100 mm VAS by marking a vertical line at the appropriate position on the scale between 0 (no pain) and 100 (most severe pain), which corresponded to the magnitude of their pain.
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
units on a scale
  General Health VAS: Week 4 (N= 473) | -20.20 (22.22)
  General Health VAS: Week 8 (N= 473) | -25.17 (24.59)
  General Health VAS: Week 16 (N= 473) | -32.54 (24.89)
  General Health VAS: Week 24 (N= 473) | -40.67 (26.28)
  Pain VAS: Week 4 (N= 473) | -24.07 (22.56)
  Pain VAS: Week 8 (N= 473) | -28.55 (24.08)
  Pain VAS: Week 16 (N= 473) | -35.20 (24.81)
  Pain VAS: Week 24 (N= 473) | -42.49 (26.05)

27. Secondary Outcome: Change in the Subject General Health VAS and Pain VAS at Each Visit During Period 2
Description: Participants were asked to answer the question "In general how would you rate your health over the last 2-3 weeks?" by marking a vertical line at the appropriate position through the 100 mm VAS. The length on the line was measured from the left (in mm). For Pain VAS, participants assessed the severity of their arthritis pain during the last 2 to 3 days using a 100 mm VAS by marking a vertical line at the appropriate position on the scale between 0 (no pain) and 100 (most severe pain), which corresponded to the magnitude of their pain.
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
units on a scale
  General Health VAS: Week 24 | -46.66 (24.72) | -47.53 (20.21)
  General Health VAS: Week 28 | -41.31 (27.01) | -34.95 (28.95)
  General Health VAS: Week 36 | -39.84 (26.56) | -30.74 (29.79)
  General Health VAS: Week 44 | -39.82 (27.61) | -30.10 (29.88)
  General Health VAS: Week 52 | -39.81 (28.16) | -29.67 (29.21)
  Pain VAS: Week 24 | -46.61 (24.33) | -49.69 (20.64)
  Pain VAS: Week 28 | -43.30 (26.34) | -38.17 (29.24)
  Pain VAS: Week 36 | -41.42 (27.01) | -34.00 (30.30)
  Pain VAS: Week 44 | -41.21 (28.01) | -33.07 (29.46)
  Pain VAS: Week 52 | -40.95 (28.61) | -32.91 (29.26)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; General Health VAS: Week 28; Test type: Superiority or Other; p = 0.078, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.21, 95% CI 2-sided [-8.91 to 0.48]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; General Health VAS: Week 36; Test type: Superiority or Other; p = 0.003, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.54, 95% CI 2-sided [-12.49 to -2.59]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; General Health VAS: Week 44; Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.19, 95% CI 2-sided [-13.20 to -3.18]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; General Health VAS: Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.60, 95% CI 2-sided [-13.64 to -3.55]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; Pain VAS: Week 28; Test type: Superiority or Other; p = 0.017, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.91, 95% CI 2-sided [-10.75 to -1.06]
Statistical Analysis 6: Comparison: Etanercept vs Placebo; Pain VAS: Week 36; Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.60, 95% CI 2-sided [-13.85 to -3.34]
Statistical Analysis 7: Comparison: Etanercept vs Placebo; Pain VAS: Week 44; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.49, 95% CI 2-sided [-14.72 to -4.26]
Statistical Analysis 8: Comparison: Etanercept vs Placebo; Pain VAS: Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -9.29, 95% CI 2-sided [-14.60 to -3.99]

28. Secondary Outcome: Change in CRP and ESR at Each Visit During Period 1
Description: as for outcome 7
Time Frame: Baseline, Weeks 4, 8, 16 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-Label Treatment
Number analyzed (Participants) | 478
units on a scale
  CRP: Week 4 (N= 465) | -14.07 (25.30)
  CRP: Week 8 (N= 471) | -14.43 (23.51)
  CRP: Week 16 (N= 472) | -14.71 (27.32)
  CRP: Week 24 (N= 472) | -14.51 (27.64)
  ESR: Week 4 (N= 473) | -17.32 (19.44)
  ESR: Week 8 (N= 473) | -19.28 (21.62)
  ESR: Week 16 (N= 473) | -21.10 (24.20)
  ESR: Week 24 (N= 473) | -26.77 (26.19)

29. Secondary Outcome: Change in CRP and ESR at Each Visit During Period 2
Description: as for outcome 7
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 163 | 168
units on a scale
  CRP: Week 24 (N= 161, 168) | -16.92 (28.64) | -14.47 (21.59)
  CRP: Week 28 (N= 160, 166) | -15.94 (28.52) | -8.59 (25.46)
  CRP: Week 36 (N= 162, 167) | -15.56 (31.36) | -7.45 (25.55)
  CRP: Week 44 (N= 162, 167) | -16.47 (30.09) | -6.72 (26.32)
  CRP: Week 52 (N= 162, 167) | -16.29 (30.74) | -7.07 (26.76)
  ESR: Week 24 (N= 163, 168) | -31.52 (22.55) | -31.02 (24.24)
  ESR: Week 28 (N= 163, 168) | -26.96 (23.04) | -20.28 (23.68)
  ESR: Week 36 (N= 163, 168) | -26.10 (24.17) | -16.94 (23.08)
  ESR: Week 44 (N= 163, 168) | -24.39 (22.99) | -16.14 (23.10)
  ESR: Week 52 (N= 163, 168) | -23.56 (21.88) | -16.27 (22.65)
Statistical Analysis 1: Comparison: Etanercept vs Placebo; CRP: Week 28; Test type: Superiority or Other; p = 0.014, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.22, 95% CI 2-sided [-9.39 to -1.05]
Statistical Analysis 2: Comparison: Etanercept vs Placebo; CRP: Week 36; Test type: Superiority or Other; p = 0.011, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.27, 95% CI 2-sided [-11.09 to -1.46]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; CRP: Week 44; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.75, 95% CI 2-sided [-12.06 to -3.44]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; CRP: Week 52; Test type: Superiority or Other; p = 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.16, 95% CI 2-sided [-11.48 to -2.85]
Statistical Analysis 5: Comparison: Etanercept vs Placebo; ESR: Week 28; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.86, 95% CI 2-sided [-9.23 to -2.49]
Statistical Analysis 6: Comparison: Etanercept vs Placebo; ESR: Week 36; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.69, 95% CI 2-sided [-12.33 to -5.05]
Statistical Analysis 7: Comparison: Etanercept vs Placebo; ESR: Week 44; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.59, 95% CI 2-sided [-11.38 to -3.80]
Statistical Analysis 8: Comparison: Etanercept vs Placebo; ESR: Week 52; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.32, 95% CI 2-sided [-10.03 to -2.60]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent to 28 days after the last dose of study medication through the last participant's visit.
Description: The Open Label Safety Population is defined as all participants who had at least one dose of open label study drug during Period 1. The Double Blind Safety Population is defined as all randomized participants who had at least one dose of study drug during period 2.
Groups:
- Open-Label Treatment: Participants in open-label treatment received ETN 50 mg with MTX (with or without other DMARDs).
Arm/Group | Open-Label Treatment | Etanercept | Placebo
Serious Adverse Events (participants affected / at risk) | 13/489 | 0/167 | 7/176
Other Adverse Events (participants affected / at risk) | 26/489 | 4/167 | 9/176
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Treatment (N=489) | Etanercept (N=167) | Placebo (N=176)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Extradural abscess (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Salmonella sepsis (Infections and infestations) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label Treatment (N=489) | Etanercept (N=167) | Placebo (N=176)
Upper respiratory tract infection (Infections and infestations) | 26 (28) | 4 (4) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.